CLINICAL TRIAL: NCT04113291
Title: Randomized Controlled Pilot Trial of Dietary Approached to Stop Hypertension (DASH) Feeding in Older Low Socioeconomic Adults Without Heart Failure
Brief Title: Randomized Controlled Pilot Trial of DASH Feeding in Older Low Socioeconomic Adults Without Heart Failure
Acronym: DASHF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DASHF-PRE
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
Keywords: DASH Diet; Low socioeconomic status; HFPEF
MeSH Terms: conditions — Heart Failure | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH diet group (Experimental): Participants randomized to receive the DASH diet will be prescribed an isocaloric DASH diet using meals (lunch, dinner, snacks) prepared by a Clinical Research Metabolic Kitchen under the direction of a registered dietician. Participants will prepare their own breakfast from a menu. The subjects will be instructed to drink no more than three caffeinated beverages and no more than two alcoholic beverages per day.
  Interventions: Other: DASH Diet
- Attention Control Group (Active Comparator): Participants randomized to attention control will continue their usual diet, but they will be instructed to limit their sodium intake to 2300 mg/day. They will be requested and voluntarily agree to not make additional diet or exercise changes during the 12-week study.
  Interventions: Other: Usual diet

INTERVENTIONS:
Other: DASH Diet — 12 Weeks of isocaloric DASH diet <2300 mg Na/day using meals (lunch, dinner, snacks) prepared by the Wake Forest Clinical Research Metabolic Kitchen under the direction of a registered dietician (RD). Participants will prepare their own breakfast from a menu.The subjects will be instructed to drink no more than three caffeinated beverages and no more than two alcoholic beverages per day.
  Other Names: Dietary Approaches to Stop Hypertension
  Arms: DASH diet group
Other: Usual diet — 12 weeks usual diet <2300 mg Na/day
  Arms: Attention Control Group

SUMMARY:
This is a study of the DASH diet (Dietary Approaches to Stop Hypertension) in the exploration of effective strategies for Heart failure (HF) with preserved ejection fraction (HFPEF) prevention.

DETAILED DESCRIPTION:
This is a feasibility pilot, randomized clinical trial (RCT), DASH diet feeding trial in 40 older adults. It will also elicit trends in left ventricular remodeling and pathophysiology. This trial investigates the feasibility of performing a DASH diet RCT intervention in HFPEF prevention in older adults of low socioeconomic status (LSES).

ELIGIBILITY:
Inclusion Criteria:

* Participants will have an education level of less than college as a surrogate marker of LSES.

Exclusion Criteria:

* Participants should not have a diagnosis of heart failure or loop diuretics on their medication list in the EHR or symptoms of dyspnea, edema (assessed via questionnaire)
* poorly controlled diabetes mellitus ( HBA 1c >9%)
* or uncontrolled hypertension ( SBP>180, DBP>110)
* cardiovascular event (MI, stroke, HF, angina, atrial fibrillation) within the previous six months
* chronic diseases that might interfere with participation (dementia, schizophrenia, dialysis or transplant recipient patients)
* body-mass index (the weight in kilograms divided by the square of the height in meters) of more than 35

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of enrolled participants per week | Up to week 12
Proportion of participants that adhere to the to intervention | Up to week 12
Number participants that were retained in the trial | Up to week 12

SECONDARY OUTCOMES:
Proportion of participants that adhere to the diet | Up to week 12

OTHER OUTCOMES:
Weight | Baseline
  Weight (kilograms)
Weight | After intervention, Week 12
  Weight (kilograms)
Waist circumference | Baseline
  Waist circumference (cm)
Waist circumference | After intervention, Week 12
  Waist circumference (cm)
Body mass Index (BMI) | Baseline
Body mass Index (BMI) | After intervention, Week 12
Systolic Blood Pressure | Baseline
Systolic Blood Pressure | After intervention, Week 12
Diastolic Blood Pressure | Baseline
Diastolic Blood Pressure | After intervention, Week 12
Total Cholesterol | Baseline
LDL Cholesterol | Baseline
HDL Cholesterol | Baseline
serum creatinine | Baseline
Total Cholesterol | After intervention, Week 12
LDL Cholesterol | After intervention, Week 12
HDL Cholesterol | After intervention, Week 12
Serum creatinine | After intervention, Week 12
Left Ventricle mass | Baseline
  Doppler-echocardiograms
Left Ventricle mass | After intervention, Week 12
  Doppler-echocardiograms
Left atrial volume | Baseline
  Doppler-echocardiograms
Left atrial volume | After intervention, Week 12
  Doppler-echocardiograms
Doppler echocardiogram velocity ratio | Baseline
Doppler echocardiogram velocity ratio | After intervention, Week 12
CRP | Baseline
  Inflammatory marker
IL6 | Baseline
  Inflammatory marker
TNF alpha | Baseline
  Inflammatory marker
CRP | After intervention, Week 12
  Inflammatory marker
IL6 | After intervention, Week 12
  Inflammatory marker
TNF alpha | After intervention, Week 12
  Inflammatory marker
6- minute walk test | Baseline
  Exercise capacity. 6- minute walk test (6 MWT) by the method of Guyatt 43. Percent predicted for age and gender.
6- minute walk test | After intervention, Week 12
  Exercise capacity. 6- minute walk test (6 MWT) by the method of Guyatt 43. Percent predicted for age and gender.
Plasma nitrate | Baseline
Plasma nitrate | After intervention, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Campos, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No